CLINICAL TRIAL: NCT01616862
Title: The Carrier Rates of Pseudomonas Aeruginosa in Family Members of Children With Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Zafer Soultan (Other)
Responsible Party: Sponsor-Investigator, Zafer Soultan, Associate professor, State University of New York - Upstate Medical University
Organization: State University of New York - Upstate Medical University (Other)
Other Study IDs: 274342
Record Dates: First submitted 2012-01-09; First posted 2012-06-12 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Pseudomonas Aeruginosa; Cystic Fibrosis
Keywords: Pseudomonas aeruginosa; cystic fibrosis
MeSH Terms: conditions — Pseudomonas Infections; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parents of PA positive CF children: parents of children with cystic fibrosis who are positive for Pseudomonas aeruginosa
- parents of Pa negative CF children: parents of children with cystic fibrosis who are negative for pseudomonas aeruginosa

SUMMARY:
Pseudomonas aeruginosa (Pa) is the bacterium that causes one of the most consequential lung infections in people with CF. Many young children do not have Pa in their lungs but will become infected as they get older. The investigators want to learn more about how Pa is passed from person to person, especially to someone with Cystic Fibrosis (CF).

DETAILED DESCRIPTION:
People with CF (cystic fibrosis) often have lung infections which occur repeatedly or worsen over time. The lung infections are most often caused by bacteria. Pseudomonas aeruginosa (Pa) is the bacterium that causes one of the most consequential lung infections in people with CF. Many young children do not have Pa in their lungs but will become infected as they get older. The investigators want to learn more about how Pa is passed from person to person, especially to someone with CF. The respiratory secretions of someone colonized with Pa can transmit or pass on the bacterium. The bacterium can be passed through direct contact by two individuals kissing or touching hands. Another way to pass Pa is by indirect contact such as touching an object like an eating utensil or drinking glass that has been used by someone with Pa.

There are many unanswered questions about Pa lung infections in people with CF. For example, it is not known why some people with CF develop Pa lung infections earlier than others. Nor is it known why it is difficult to eradicate Pa in some children and why some children's condition to deteriorate quicker than other after becoming infected with Pa.

Biological parents of children with CF are carriers of one CF causing gene mutation. It is also possible that they are carriers of additional, but milder, CF-related gene mutations. It is possible that the carrier status of the parents of CF children place them at risk of acquiring and carrying Pa in their lungs.

Biological parents of children who have CF will be asked to participate. This study plans to assess the frequency of Pa in biological parents and to correlate the clinical and microbiological status of CF children with PA carrier rates of their parents.

Parents will be asked to complete questionnaires at one routine, clinic visit, have nasal and throat cultures collected during their child's routine scheduled visit and again 3-4 months later (at another routine visit). The investigators are also asking permission to review the medical records of their child with CF.

ELIGIBILITY:
Inclusion Criteria:

* Biological parents of children with CF will be invited to participate and included if their children meet the following criteria:

  * children's age is more than 5 years and less than 20 years of age.

Exclusion Criteria:

* Biological parents of children younger than 5 years of age or older than 20 years of age.
* Step parents.

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Biological parents of children with cystic fibrosis who are treated at Upstate Medical University. Children's age is more than 5 yrs and less than 20 yrs.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Primary objective: the incidence of Pseudomonas aeruginosa colonization in the upper respiratory tract of parents of children with CF. | 6 months
  Collection of nasal and oropharyngeal swabs will be obtained from parents living with patients at enrollment and after 3 months.
Primary objective: the incidence of Pseudomonas aeruginosa colonization in the upper respiratory tract of parents of children with CF. | Day 0
  Collection of nasal and oropharyngeal swabs will be obtained from parents living with patients at enrollment and after 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Zafer Soultan, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

REFERENCES:
- [Background] Microbiology and infectious disease in cystic fibrosis. Clinical Practice Guidelines for Cystic fibrosis; Cystic Fibrosis Foundation; Appendix V111, Volume V, Section I May 17-18, 1994
- [Background] Kerem E, Rave-Harel N, Augarten A, Madgar I, Nissim-Rafinia M, Yahav Y, Goshen R, Bentur L, Rivlin J, Aviram M, Genem A, Chiba-Falek O, Kraemer MR, Simon A, Branski D, Kerem B. A cystic fibrosis transmembrane conductance regulator splice variant with partial penetrance associated with variable cystic fibrosis presentations. Am J Respir Crit Care Med. 1997 Jun;155(6):1914-20. doi: 10.1164/ajrccm.155.6.9196095.
- [Background] Joel Moss form Pulmonary-Critical Care Medicine Branch, NHLBI, National Institutes of Health, Bethesda, Maryland, presented data stating that carriers of a CFTR gene mutations can be colonized by Pseudomonas aeruginoa. The data presented at The American Thoracic Society International Conference - 2005; in a seminar on Pseudomonas aeruginosa.
- [Background] HUANG NN, SHEN KT. Staphylococcal carrier rates of patients with cystic fibrosis and of members of their families. J Pediatr. 1963 Jan;62:36-43. doi: 10.1016/s0022-3476(63)80068-2. No abstract available. PMID 13955349